CLINICAL TRIAL: NCT01009398
Title: Radiological Evaluation of Thoracic Paravertebral Catheters: A Prospective Clinical Trial
Brief Title: Thoracic Paravertebral Catheters
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Cédric Luyet, M.D., University Hospital and Universtiy of Bern, Department of Anaesthesiology and Pain Therapy
Other Study IDs: 167/09
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Thoracic Paravertebral Block
Keywords: Anesthesia and Analgesia; Regional anesthesia; Thoracic Paravertebral block; Catheter location
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fluoroscopic examination — Localisation of the paravertebral catheter tip and documentation of the spread of contrast dye injected through the catheters by fluoroscopic examination

SUMMARY:
Thoracic operations are known to be painful and requiring an adequate postoperative pain therapy. A well documented technique to achieve postoperative analgesia is the use of paravertebral catheters. Theoretically the thoracic paravertebral block results in an unilateral thoracic anaesthesia. However, in the daily clinical practice it remains unclear whether catheters are placed correctly into the paravertebral region. The investigators' experiences with paravertebral catheters suggest that there may be many displacements of catheters since the pain control is reduced compared to epidural analgesia.

The aim of this prospective observational clinical trial is to postoperatively evaluate the exact location of paravertebral catheter placed for thoracoscopic interventions by using the classical land-mark puncture technique. After radiological detection of the catheter position, the spread and distribution of contrast dye injected through the catheters will be evaluated.

DETAILED DESCRIPTION:
Background

The paravertebral block is a regional anaesthetic technique which can be used for analgesia after thoracic, cardiac, breast surgery, upper abdominal surgery or for pain therapy. Thoracic paravertebral blockade is performed by injecting a local anaesthetic solution into the paravertebral space, which contains the thoracic nerves, their branches and the sympathetic trunk. This space is a wedge-shaped area sandwiched between the heads and necks of the ribs. The posterior wall is formed by the superior costo-transverse ligament, the antero-lateral wall is the parietal pleura with the endothoracic fascia and the medial wall is the lateral surface of the vertebral body and disc. Also medially, there is communication with the epidural space via the intervertebral foramen. It has been shown, that each space communicates inferiorly and superiorly across the heads and necks of the ribs. Thus injecting local anaesthetic in the paravertebral space should results to an analgesia corresponding to a unilateral epidural anaesthesia.

Unilateral multisegmental anaesthesia after single-shot paravertebral injection of local anaesthetics is well established. On the other hand, a variety of different studies on volunteers, patients and cadavers showed conflicting results regarding the vertical spread over several adjacent segments after paravertebral injection leading to the recommendation of some authors to use a multi-injection technique to achieve a multilevel somatic nerve blockade, specially described during breast surgery using paravertebral block alone.

Can we explain these different contradictory reports and recommendations? Available radiologic and anatomic studies show many different patterns of contrast dye spread after single shot paravertebral contrast dye injection. One study even reports different distribution of dye even after several paravertebral single shots of the same operator in the same patient. Some radiological studies report cloud-like contrast dye accumulation without significant cranio-caudal spread. This could be due to the restricted intercostal spread or to subpleural spread or even to injection of the contrast dye into the autochthonic muscles of the back.

The spread of local anesthetics (or contrast dye as substitute) is affected by nuances of differences in the needle placement because of the fine membranes like the endothoracica fascia. This might be the major problem during the insertion of catheters. The final location of catheter tip is hard to predict. Catheters might dissect during the insertion and possibly the difference is only a more medial or more lateral puncture. The placement of catheters into the paravertebral space leading to a clear cranio-caudal spread of local anaesthetics resulting in multisegmental spread of anaesthesia is the goal of a catheter for paravertebral analgesia but it seems not easy to be achieved - despite of an uncontestable clinical benefit of paravertebral catheters for pain relief.

Studies describing the exact emplacement of catheters, distribution of contrast dye and correlation of this distribution with the clinical effect after catheter placement by the classical land-mark based approach as described by Eason and Wyatt are lacking. We therefore aim to describe the different possible emplacements of the catheters, the resulting spread of contrast dye after injection through the catheters as well as the corresponding area of somatic and sympathetic block.

Objective

The aim of prospective observational clinical trial is to evaluate the exact location of paravertebral catheter placed for thoracoscopic interventions using the classic landmark approach by injecting a small amount of contrast dye (1 ml) through the catheter and subsequent fluoroscopic documentation of the catheter tip localisation. Thereafter a larger amount (20 ml) of diluted contrast dye will be injected and its spread will be documented fluoroscopically.

Methods

Once the paravertebral catheter is placed as usual after the end of surgery, 1 ml of contrast dye will be injected through the catheter. After fluoroscopic documentation of the catheter tip, further 10 ml of diluted contrast dye will be injected and its spread again documented fluoroscopically in two planes. All saved pictures, showing the catheter tip position and the contrast dye spread, will be evaluated subsequently by an independent radiologist. After these fluoroscopic examinations a test dose of Bupivacaine 0.25% mixed with Adrenaline 5 mcg/ml of 3ml will be injected through the catheter followed by an injection of 0.3ml/kg of local anaesthetics (Bupivacaine 0.25% mixed with Adrenaline 5 mcg/ml). One hour later a clinical testing of the skin area with somatic and sympathetic block provided through the paravertebral catheters will be performed and the data recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for thoracoscopic intervention
* Planned placement of paravertebral catheters

Exclusion Criteria

* Refusal to participate
* Age < 18
* Severe hepatic disfunction (Liver disease Child B or C)
* known allergies to iodinated contrast material
* Morbus Waldenström
* multiple myeloma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are scheduled for a thoracoscopic intervention with planned placement of paravertebral catheters as their standard postoperative pain treatment strategy are eligible for this prospective observational clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Exact position of the paravertebral catheter | immediately

SECONDARY OUTCOMES:
Spread of contrast dye through the catheters | immediately
Correlation of clinical effect of local anaesthetics injected through the catheters and documented spread of contrast dye | immediately

CONTACTS AND LOCATIONS:
Overall Officials: Urs Eichenberger, M.D., Study Chair — University Hospital and University of Bern, Department of Anaesthesiology and Pain therapy
Locations (1):
- University Hospital and University of Bern, Department of Anaesthesiology and Pain Therapy, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Eason MJ, Wyatt R. Paravertebral thoracic block-a reappraisal. Anaesthesia. 1979 Jul-Aug;34(7):638-42. doi: 10.1111/j.1365-2044.1979.tb06363.x. PMID 517716
- [Background] Hill SE, Keller RA, Stafford-Smith M, Grichnik K, White WD, D'Amico TA, Newman MF. Efficacy of single-dose, multilevel paravertebral nerve blockade for analgesia after thoracoscopic procedures. Anesthesiology. 2006 May;104(5):1047-53. doi: 10.1097/00000542-200605000-00022. PMID 16645458
- [Background] Luyet C, Eichenberger U, Greif R, Vogt A, Szucs Farkas Z, Moriggl B. Ultrasound-guided paravertebral puncture and placement of catheters in human cadavers: an imaging study. Br J Anaesth. 2009 Apr;102(4):534-9. doi: 10.1093/bja/aep015. Epub 2009 Feb 24. PMID 19244265